CLINICAL TRIAL: NCT06150690
Title: Study on the Function of Insulin-producing Beta Cells in the Human Pancreas
Brief Title: Study on Pancreatic Islets in Patients Undergoing (Partial) Pancreatectomy (PRECISE)
Acronym: PRECISE
Status: Recruiting | Type: Observational
Sponsor: German Diabetes Center (Other)
Collaborators: Lukas Hospital, Neuss, Germany (Unknown); Heinrich-Heine University, Duesseldorf (Other); Florence Nightingale Hospital, Düsseldorf, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: Pancreatic-Islet-Study-01
Record Dates: First submitted 2019-09-12; First posted 2023-11-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Pancreatic tissue, visceral adipose tissue and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Type 2 diabetes: Patients with type 2 diabetes undergoing (partial) pancreatectomy
  Interventions: Other: No intervention
- Type 3 diabetes: Patients with type 3 diabetes undergoing (partial) pancreatectomy
  Interventions: Other: No intervention
- Non-diabetic controls: Patients with normal glucose metabolism undergoing (partial) pancreatectomy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — The participants did not receive any study-specific intervention

SUMMARY:
The study investigates the mechanisms underlying the pathogenesis of diabetes by examining structural and functional properties of islets of Langerhans in pancreas specimen from patients undergoing (partial) pancreatectomy.

DETAILED DESCRIPTION:
The study aims at elucidating the mechanisms underlying the pathogenesis of diabetes. In particular, the study focusses on detailed analyses of morphological and functional properties of pancreatic islets/insulin-producing beta cells in order to identify diabetes-associated alterations on cellular and molecular levels. To directly address the role of the endocrine (and exocrine) pancreas in the complex process of diabetes development, the examinations are performed in samples of human pancreatic tissue. To this end, biopsy specimen of pancreas and visceral adipose tissue are collected from patients with or without diabetes who undergo (partial) pancreatectomy. The samples are analysed for morphological alterations (e.g. size and distribution of pancreatic islets and beta cells, size of adipocytes) and functional changes (e.g. gene expression patterns as assessed from beta-cell derived RNA). In addition, patient characteristics such as age and disease duration are documented and clinical data including fasting concentrations of blood glucose, insulin and free fatty acids are collected. Specific diabetes-associated alterations of pancreatic islet / beta cells are assessed by associating variables of glucose- and lipid-homeostasis with parameters of beta cell function. The expected outcomes of the study will contribute to improve our knowledge of the so far largely unknown molecular and cellular mechanisms involved in the pathogenesis of diabetes.

ELIGIBILITY:
Inclusion Criteria:

ability to give informed consent

Exclusion Criteria:

denial of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with or without diabetes who undergo (partial) pancreatectomy
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-08-21 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Glycated hemoglobin | 1 year
  Proportion of glycated HbA1c (in %) as determined from pre-operative serum samples

SECONDARY OUTCOMES:
Islet area | 1 year
  Size of pancreatic islets of Langerhans (in square micrometers) as determined by microscopic/morphometric analyses of appropriately stained thin sections of pancreatic tissue samples

CONTACTS AND LOCATIONS:
Overall Officials: Michael Roden, Prof MD, Principal Investigator — German Diabetes Center
Locations (1):
- German Diabetes Center, Düsseldorf, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Böddeker J-S, Burkart V, Strassburger K, Goretzki P, Knoefel W-T, Möbius C, Bug R, Hinsch N, Esposito I, Gerharz CD, Roden M, Müssig K. Diabetes in Patients with Pancreatic Cancer: Relationship of Tumor Grade with Glycemic Control. Diabetes 2019; 68 (Suppl 1) DOI: https://doi.org/10.2337/db19-434-P